CLINICAL TRIAL: NCT03434795
Title: Distinction Risk of Severe Infection in Febrile Neutropenia After Chemotherapy: a Multicenter Validation of Clinical Decision Rule
Brief Title: Distinction Risk of Severe Infection in Febrile Neutropenia After Chemotherapy
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government); Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2011_40; 912180 (Other: CNIL number); 12-272 (Other: CCTIRS number)
Record Dates: First submitted 2018-01-18; First posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Febrile Neutropenia, Rule of Clinical Decision, Chemotherapy
MeSH Terms: conditions — Febrile Neutropenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluate the reproducibility and validate a posteriori a new rule of clinical decision on a multi-center population of children with a post-chemotherapy febrile neutropenia

ELIGIBILITY:
Inclusion Criteria:

* Child aged 1 to 18 years
* Child with hematology or cancer
* Child with a febrile neutropenia post-chemotherapy
* Child with social security
* No opposition from the child and/or parents, in case of absence, the holder of the parental authority present, can consent, alone, to the participation of the unemancipated minor.

Exclusion Criteria:

* Febrile neutropenia at diagnosis of tumor disease
* Child with palliative care
* Child having had a hematopoietic stem cell allo-graft in the preceding year
* Febrile neutropenia immediately post auto-transplant
* Antibiotherapy prior to admission
* Initial care in a non-investigative center.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patient with hematology or cancer who consults for febrile neutropenia post-chemotherapy
Sampling Method: Probability Sample
Enrollment: 1900 (Actual)
Dates: Start 2012-05; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Blood culture | On average between 5 days and 1 month
  Presence or not of bacteriemia
Positive bacterial culture from a normally sterile site | on average between 5 days and 1 month
  Presence or not of bacterial infection
microbiological culture | On average between 5 days and 1 month
  Presence or not of focal infection at high risk of dissemination was defined as any local infection with or without microbiological documentation into a normally sterile site, with significant risk of loco-regional or systemic spread
Fungal culture | On average between 5 days and 1 month
  Presence or not of fungal infection is referred to a proven, probable, or possible fungal infection as defined by the IFICG ot the EORTC

CONTACTS AND LOCATIONS:
Overall Officials: François Dubos, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Jeanne de Flandre - CHRU de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Delebarre M, Gonzales F, Behal H, Tiphaine A, Sudour-Bonnange H, Lutun A, Abbou S, Pertuisel S, Thouvenin-Doulet S, Pellier I, Mansuy L, Piguet C, Paillard C, Blanc L, Thebaud E, Plantaz D, Blouin P, Schneider P, Guillaumat C, Simon P, Domenech C, Pacquement H, Le Meignen M, Pluchart C, Verite C, Plat G, Martinot A, Duhamel A, Dubos F. Decision-tree derivation and external validation of a new clinical decision rule (DISCERN-FN) to predict the risk of severe infection during febrile neutropenia in children treated for cancer. Lancet Child Adolesc Health. 2022 Apr;6(4):260-268. doi: 10.1016/S2352-4642(21)00337-0. Epub 2021 Dec 3. PMID 34871572